CLINICAL TRIAL: NCT05190861
Title: Evaluation of Droplet Digital PCR Rapid Detection Method and Precise Diagnosis and Treatment for Suspected Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PROGRESS
Record Dates: First submitted 2021-11-25; First posted 2022-01-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2022-01

CONDITIONS: Sepsis; Septic Shock
Keywords: Digital Droplet PCR; Etiology Diagnose
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Blood Culture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- droplet digital PCR method (Experimental): Pathogen detection by droplet digital PCR method as an adjunct to traditional microbiological assessments including blood culture
  Interventions: Diagnostic Test: droplet digital PCR method
- blood culture only (Active Comparator): Pathogen detection by microbiological assessments including blood culture
  Interventions: Diagnostic Test: blood culture

INTERVENTIONS:
Diagnostic Test: droplet digital PCR method — The droplet digital PCR method can detect nucleic acids from the most common pathogens (approximately 90%) responsible for BSIs according to Chinet2020 and takes about 4 hours to perform, reporting within the first 24h of suspected sepsis/septic shock.
  Arms: droplet digital PCR method
Diagnostic Test: blood culture — Blood culture is a conventional microbiological method of pathogen detection. Results from blood cultures are usually not available until 24 to 72 hours after sampling.
  Arms: blood culture only

SUMMARY:
Sepsis is a significant public health concern worldwide, with high morbidity and mortality. With regard to a targeted antimicrobial treatment strategy, the earliest possible pathogen detection is of crucial importance. Until now, culture-based detection methods represent the diagnostic gold standard, although they are characterized by numerous limitations. Culture-independent molecular diagnostic procedures may represent a promising alternative. In particular, droplet digital PCR (ddPCR) is a novel one-step PCR assay that achieves higher accuracy and sensitivity in detecting causing pathogens in patients with bloodstream infections.

ELIGIBILITY:
Inclusion Criteria:

1.18 years or older

2.Meet 2 of 4 sepsis criteria

1. Temperature > 38C or < 36C
2. Heart rate > 90 bpm
3. Respiratory rate >20 or PaCO2 <32mmHg
4. WBC >12000/µL or < 4000/µL or > 10% bands

   3.Hospitalized patients who have a diagnostic blood culture ordered as standard of care for suspected sepsis

   4.Informed Consent by patient or legal representative.

   Exclusion Criteria:
   1. Refusal to participate in the study or Failure to comply with treatment or follow-up time
   2. Known breastfeeding or pregnancy
   3. The researcher believes that there are any conditions (social or medical) that allow subjects to participate is unsafe. For example, severe anemia or high risk of bleeding,etc., which are not suitable for taking peripheral blood for testing
   4. Participating in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1032 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Up to 96 hours post blood collection
  The primary endpoint of estimated sensitivity will be determined by comparing positive blood culture results with the concomitantly collected ddPCR results from the prospective clinical specimens.
Specificity | Up to 96 hours post blood collection
  The primary endpoint of estimated specificity will be determined by comparing negative blood culture results with the concomitantly collected ddPCR results from the prospective clinical specimens.

SECONDARY OUTCOMES:
Time to the change to the targeted antimicrobial therapy | At time point of change to the targeted antimicrobial therapy, up to 96 hours post blood collection
Number of patients with targeted antimicrobial therapy | Up to the end of study participation, an average of 1 year
Time to identification of a potential pathogen | At time point of identification of a potential pathogen, up to 96 hours post blood collection
Duration of antimicrobials | Up to the end of study participation, an average of 1 year
Change in condition severity | Up to the end of study participation, an average of 1 year
  The sequential organ failure assessment score (SOFA score), previously known as the sepsis-related organ failure assessment score, higher scores mean worse outcome.
Days in intensive care unit (ICU) | Up to the end of study participation, an average of 1 year
Ventilation duration in ICU (hours) | Up to the end of study participation, an average of 1 year
Days in hospital (from study inclusion) | Up to the end of study participation, an average of 1 year
All-cause death | Up to the end of study participation, an average of 1 year
Treatment costs | Up to the end of study participation, an average of 1 year
Quality of life of survivors after being discharged | Up to the end of study participation, an average of 1 year
  EQ-5D, a standardised measure of health-related quality of life developed by the EuroQol Group.The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. The number of levels in these dimensions is 5 in the EQ-5D-5L. Higher levels mean worse health states.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Nanjing Hospital of Chinese Medicine Affiliated to Nanjing University of Chinese Medicine, Nanjing, Jiangsu
  - Wuxi No.5 People's Hospital, Wuxi, Jiangsu
  - Xinhua Hospital Affliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Minhang Branch of Ruijin Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Rui'an People's Hospital, Rui’an, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao Y, Lin K, Zhang H, Zhang Y, Li S, Zhang S, Zhang W, Zhou A, Zhuang Y, Chen J, Wu C, Zhou W, He X, Yue Q, Zhang M, Huang Y, Li L, Hong L, Cai F, Huang L, Ruan Z, Xu S, Zhang Y, Chen X, Chen J, Ye Y, Bian T, Li J, Yin J, Li X, Jiang L, Lei C, Liu J, Zhang Y, Jin J, Ai J, Pan J, Zhang W. Prognostic value of poly-microorganisms detected by droplet digital PCR and pathogen load kinetics in sepsis patients: a multi-center prospective cohort study. Microbiol Spectr. 2024 May 2;12(5):e0255823. doi: 10.1128/spectrum.02558-23. Epub 2024 Mar 25. PMID 38526296
- [Derived] Zhao Y, Lin K, Zhang H, Yuan G, Zhang Y, Pan J, Hong L, Huang Y, Ye Y, Huang L, Chen X, Liu J, Li X, He X, Yue Q, Zhang H, Zhou A, Zhuang Y, Chen J, Wu C, Zhou W, Cai F, Zhang S, Li L, Li S, Bian T, Li J, Yin J, Ruan Z, Xu S, Zhang Y, Chen J, Zhang Y, Han J, Su T, Tu F, Jiang L, Lei C, Du Q, Ai J, Zhang W. Evaluation of droplet digital PCR rapid detection method and precise diagnosis and treatment for suspected sepsis (PROGRESS): a study protocol for a multi-center pragmatic randomized controlled trial. BMC Infect Dis. 2022 Jul 19;22(1):630. doi: 10.1186/s12879-022-07557-2. PMID 35854212